CLINICAL TRIAL: NCT03620461
Title: Epidemiological, Observational, Retrospective and Multicenter Study to Evaluate the Characteristics of Treatment With Gemcitabine and Nab-paclitaxel in Patients With Metastatic Pancreatic Adenocarcinoma Treated in the First Line in Routine Clinical Practice. ANICE-PaC Study
Brief Title: Gemcitabine and Nabpaclitaxel in Metastatic Pancreatic Carcinoma.
Acronym: ANICE-PaC
Status: Completed | Type: Observational
Sponsor: Galician Research Group on Digestive Tumors (Other)
Responsible Party: Sponsor
Other Study IDs: gitud
Record Dates: First submitted 2018-06-04; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: metastatic pancreatic cancer; real world data; gemcitabine; nabpaclitaxel; efficacy; safety
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Gemcitabine - nabpaclitaxel — efficacy and safety

SUMMARY:
Retrospective, multicenter study including pts with metastatic pancreatic cancer who started first-line treatment with napaclitaxel plus Gemcitabine between December 2013 and June 2015 according to the routine practice. Overall survival (OS) and progression-free survival (PFS) were assessed for the total sample and the exploratory subgroups based on treatment and clinical characteristics of the study pts.

DETAILED DESCRIPTION:
This observational, retrospective, multicenter study included patients with metastatic pancreatic adenocarcinoma (either recurrent or de novo) from 20 Spanish hospitals, who started first-line chemotherapy with nab-paclitaxel (Abraxane®, Celgene Europe Limited) plus gemcitabine between December 2013 and June 2015 according to routine clinical practice. The record included all adult patients (i.e., aged ≥ 18 years) with measurable metastatic disease at baseline in at least one dimension of the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1,[15] who received at least one dose of combined treatment with nab-paclitaxel plus gemcitabine. Data were retrieved from patients' medical records and lasted until death or the closure of the database on 16 March 2017. All patients signed the corresponding informed consent for their clinical data being used in this study, which was conducted in accordance with the local personal data protection law (LOPD 15/1999). The study protocol was approved by the local independent ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed pancreatic adenocarcinoma or poorly differentiated carcinoma that is metastatic to distant sites.
* Other histologies such as neuroendocrine and acinar cell carcinoma are excluded.
* No prior chemotherapy for metastatic pancreatic cancer.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Age greater than or equal to 18 years.
* Patient has signed a Patient Informed Consent Form.
* Patients should have received at least one cycle of gemcitabine and nabpaclitaxel

Exclusion Criteria:

* less than one cycle of gemcitabine/nabpaclitaxel administrated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (i.e., aged ≥ 18 years) with measurable metastatic disease at baseline in at least one dimension of the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1,[15] who received at least one dose of combined treatment with nab-paclitaxel plus gemcitabine
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 2 years
  Evaluate overall survival (OS) in patients with metastatic pancreatic cancer receiving gemcitabine and nab-paclitaxel
progression free survival | 2 years
  Evaluate progression free survival (PFS) in patients with metastatic pancreatic cancer receiving gemcitabine and nab-paclitaxel
Assess adverse events (per CTCAE v4.0 criteria) | 2 years
  Assess the adverse events (per CTCAE v4.0 criteria) associated with the use of gemcitabine and nab-paclitaxel in real world setting.

IPD SHARING:
Plan to Share IPD: Undecided